CLINICAL TRIAL: NCT02435537
Title: Safety and Efficacy of Dexmedetomidine Addition to Intrathecal Morphine for Postoperative Analgesia in Cancer Patients Undergoing Major Abdominal Surgery
Brief Title: Combined Intrathecal Morphine and Dexmedetomidine Analgesia
Acronym: ITMandDEX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Fares, Professor in Anesthesia and intensive care department, South Egypt Cancer institute, Assiut university, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IORG0006563/reference. no. 64
Record Dates: First submitted 2015-04-26; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Pain
Keywords: analgesia; intrathecal; opioids; morphine; dexmedetomidine
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexmedetomidine; Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intrathecal Bupivacaine (Active Comparator): intrathecal injection of 10 mg hyperbaric bupivacaine 0.5% in 2 ml volume and 1ml of saline 0.9%
  Interventions: Drug: Bupivacaine
- Intrathecal Morphine (Active Comparator): intrathecal injection of 10mg bupivacaine 0.5% in 2ml volume intrathecal injection of 0.5 mg morphine in 1ml volume
  Interventions: Drug: Bupivacaine; Drug: Morphine
- Intrathecal Morphine-Dex (Active Comparator): intrathecal 10mg bupivacaine 0.5% in 2 ml volume intrathecal 0.5 mg morphine intrathecal 5 µg of dexmedetomidine in 1ml volume .
  Interventions: Drug: Dexmedetomidine (Precedex); Drug: Bupivacaine; Drug: Morphine

INTERVENTIONS:
Drug: Dexmedetomidine (Precedex) — intrathecal administration
  Other Names: Precedex
  Arms: Intrathecal Morphine-Dex
Drug: Bupivacaine — intrathecal 10 mg bupivacaine
  Other Names: Buvicaine
Drug: Morphine — intrathecal 0.5mg morphine
  Other Names: morphine sulphate
  Arms: Intrathecal Morphine; Intrathecal Morphine-Dex

SUMMARY:
The current study investigated the effect of adding dexmedetomidine to intrathecal morphine for postoperative analgesia in cancer patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
Opioids, administered intrathecal or epidural, are widely used for postoperative, and chronic nociceptive pain secondary to cancers. Intrathecal injection of morphine to provide postoperative analgesia during the initial 24 h after operation is a widely used technique.The Human studies on the antinociceptive effects of co-administrated intrathecal morphine and dexmedetomidine in postoperative pain are still lacking. In this study, the investigators aimed to compare the synergistic interaction and side-effects of combined intrathecal morphine and dexmedetomidine with either drug alone for postoperative analgesia in cancer patients undergoing major abdominal surgery. Patients were randomly allocated into three groups of 30 patients each to receive either; hyperbaric bupivacaine 0.5% (Group I/Bupivacaine Group), bupivacaine and 0.5 mg morphine (Group II/Morphine Group), bupivacaine and 0.5 mg morphine plus 5 µg of dexmedetomidine (Group III/Morphine-DEX Group). The assigned drugs were dissolved in 1ml physiological saline and administered intrathecal with bupivacaine before induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

- major abdominal cancer surgery (e.g. hemi-colectomy or cystectomy)

Exclusion Criteria:

* known allergy to study drugs
* Significant cardiac, respiratory, renal or hepatic disease.
* 2nd or 3rd degree heart block.
* Coagulation disorders.
* Low back pain or other back problems.
* Drug or alcohol abuse.
* BMI>30kg\m2.
* Psychiatric illnesses that would interfere with perception and assessment of pain.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
total dose of intravenous PCA morphine consumption in the first 48 h postoperative | 48 hours
  Calculating the cumulative intravenous PCA morphine dose

SECONDARY OUTCOMES:
Noninvasive blood pressure | 48 hours
  non invasive systolic and diastolic blood pressure intra-operative and postoperative in the 6th, 12th, 18th, 24th, 36th, and 48th h postoperative.
Heart rate | 48 hours
  non invasive assessment of heart rate in the 6th, 12th, 18th, 24th, 36th, and 48th postoperative. intraoperative and postoperative
peripheral arterial oxygen saturation | 48 hours
  assessment of pulse oximetry intraoperative and in the 6th, 12th, 18th, 24th, 36th, and 48th h postoperative
postoperative VAS scores | 48 hours
  assessment of pain scores on admission to surgical intensive care unit and in the 6th, 12th, 18th, 24th, 36th, and 48th h postoperative.
time to first request for analgesia | 48hours
  measuring the time in hours of first request for intravenous PCA morphine

CONTACTS AND LOCATIONS:
Overall Officials: Saher AB Mohamed, MD, Study Director — Assisstant professor in Anesthesia and intensive care department, South Egypt Cancer institute, Assiut university, Egypt; Hala s Abdel-Ghaffar, MD, Study Director — Assisstant professor in Anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt.

REFERENCES:
- [Derived] Abdel-Ghaffar HS, Mohamed SA, Fares KM. Combined Intrathecal Morphine and Dexmedetomidine for Postoperative Analgesia in Patients Undergoing Major Abdominal Cancer Surgery. Pain Med. 2016 Nov;17(11):2109-2118. doi: 10.1093/pm/pnw031. Epub 2016 Mar 21. PMID 27002003